CLINICAL TRIAL: NCT07387965
Title: A Brief Psychoeducation Intervention to Address Cannabis Use Amongst Patients Seeking Eating Disorder Treatment: A Single Blind Randomized Control Trial
Brief Title: A Brief Cannabis Use Psychoeducation Intervention for Eating Disorder Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Sarah McComb, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18846
Record Dates: First submitted 2026-01-13; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Eating Disorders; Cannabis Use
Keywords: single blind; single blind randomized control trial; randomized control trial; eating disorders; cannabis use; psychoeducation; brief intervention; marijuana; cannabis; binge eating disorder; anorexia nervosa; bulimia nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Marijuana Abuse; Binge-Eating Disorder; Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabis psychoeducation intervention (Experimental): Brief psychoeducation will be provided to eating disorder patients seeking treatment regarding the impact of cannabis use on comorbid mental health conditions, sleep, gastrointestinal symptoms, eating disorder symptoms, and eating disorder treatment outcomes.
  Interventions: Other: Psychoeducation about risks of cannabis use
- Psychoeducation control condition (Placebo Comparator): Brief psychoeducation will be provided to eating disorder patients seeking treatment regarding the impact of poor sleep on mental health outcomes and appropriate sleep hygiene habits.
  Interventions: Other: Placebo control: Sleep hygiene psychoeducation

INTERVENTIONS:
Other: Psychoeducation about risks of cannabis use — This intervention will provide psychoeducation to eating disorder patients about the risks of using cannabis on mood, anxiety, sleep, substance use, gastrointestinal symptoms, eating disorder symptoms, and eating disorder treatment outcomes.
  Arms: Cannabis psychoeducation intervention
Other: Placebo control: Sleep hygiene psychoeducation — Eating disorder patients in the control condition will receive psychoeducation about impacts of poor sleep on mental health and eating disorder treatment outcomes, and strategies to improve sleep hygiene.
  Arms: Psychoeducation control condition

SUMMARY:
The goal of this clinical trial is to learn if providing eating disorder patients with education about the consequences of cannabis (marijuana) use on mental health, gastrointestinal symptoms, eating disorder symptoms, and eating disorder treatment effectiveness increases their knowledge about the cannabis use consequences, intention to reduce cannabis use, and motivation to seek treatment for their cannabis use. The main questions this study aims to answer are:

1. Does education about consequences of cannabis use increase eating disorder patients' knowledge about the risks of cannabis use?
2. Does education about the consequences of cannabis use increase intention to reduce cannabis use and seek cannabis use treatment among those with eating disorders?
3. Does cannabis use interfere with how successful eating disorder treatment is for eating disorder patients?

All participants will receive 20 weeks of eating disorder treatment. In week 1 of treatment, participants will either be assigned to receive education about cannabis use consequences, or be assigned to a control condition where they receive education about consequences of poor sleep. Participants will be asked to complete a number of questionnaires that measure knowledge about cannabis use consequences, intention to reduce use and seek cannabis use treatment, eating disorder symptoms, and cannabis use habits. Researchers will assess how effective providing education about cannabis use consequences is on changing knowledge about cannabis use risks, intention to reduce use, and intention to seek cannabis use treatment. It will also be examined if effectiveness of eating disorder treatment is related to cannabis use habits.

ELIGIBILITY:
Inclusion Criteria:

* A patient of St. Joseph's Healthcare Hamilton Eating Disorder Program (i.e. is currently seeking eating disorders treatment)
* Participant has been diagnosed with an eating disorder
* Aged 16+
* Understands written and spoken English

Exclusion Criteria:

* Has not been diagnosed with an eating disorder
* Under the age of 17
* Does not understand written and spoken English

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2028-02-04 (Estimated); Study Completion 2028-02-04 (Estimated)

PRIMARY OUTCOMES:
Knowledge of cannabis use consequences | Will be measured at baseline (i.e. 5 minutes into Session 1 of treatment for eating disorders before cannabis psychoeducation is administered), and again at 140 minutes into Session 1 of treatment for eating disorders.
  Self-perceived knowledge about consequences of cannabis use will be measured using a 100 point visual analogue scale. Higher scores will indicate greater self-perceived knowledge about the consequences of cannabis use.
Intention to reduce cannabis use | Will be measured at baseline (i.e. 5 minutes into Session 1 of treatment for eating disorders before cannabis psychoeducation is administered), and again at 140 minutes into Session 1 of treatment for eating disorders.
  Intention to reduce personal cannabis use will be measured using a 100 point visual analogue scale. Higher scores indicate greater intention to reduce cannabis use.
Intention to seek cannabis use treatment | Will be measured at baseline (i.e. 5 minutes into Session 1 of treatment for eating disorders before cannabis psychoeducation is administered), and again at 140 minutes into Session 1 of treatment for eating disorders.
  Intention to seek cannabis use treatment will be measured using a 100 point visual analogue scale. Higher scores indicate greater intention to seek cannabis use treatment.

SECONDARY OUTCOMES:
Motivations for cannabis use | Measured at baseline (i.e. Week 1 of CBT for eating disorders) and through treatment completion (i.e. Week 20 of CBT for eating disorders).
  Motivations for cannabis use will be measured using the Marijuana Motives Questionnaire (5 subscales measuring motivations regarding enhancement, coping, conformity, expansion, and social). Responses range from 1 to 5, with higher scores indicating greater endorsement of that motivation. Subscale scores are calculated by taking the average score of subscale items.
  Motivations for cannabis use will also be measured using the Comprehensive Cannabis Motivates Questionnaire (8 subscales measuring motivations regarding food, medicinal, sleep, social, to get high, coping, conformity, creativity). Responses range from 1-5, with higher scores indicating greater endorsement of that motivation. Subscale scores are calculated by taking the average score of subscale items.
Cannabis use frequency | Weekly use will be monitored for 20 weeks using a Likert-type question. The Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use Inventory will be measured twice during Week 1 and Week 20 of CBT for eating disorders
  Will be measured weekly for 20 weeks using a Likert-type question and at Week 1 and Week 20 of CBT for eating disorders using the Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use Inventory.
Eating disorder symptoms | Administered at Week 1 (baseline) and Week 20 of CBT for eating disorders.
  Measured using the Eating Disorder Examination Questionnaire, which assesses for symptoms such as restrictive eating, binge eating, purging, exercise, and body image. This measure has 4 subscale scores (restraint, concern about eating, weight concerns, and shape concerns) and one global score. Items are answered on a scale of 0 to 6, with higher scores indicating greater eating disorder symptoms. Subscale scores are calculated by taking the average of subscale item scores. The global score is calculated by averaging the sum of the 4 subscale scores.
Impairment caused by eating disorder | Administered at Week 1 and Week 20 of CBT for eating disorders.
  Measured using the Clinical Impairment Assessment. Assesses for impairment caused by eating disorder symptoms, such as negative emotions, concentration difficulties, social impairment. Items are responded to on a scale of 0 to 3, with higher scores indicating greater impairment on that item. A total score is calculated by summing all item scores.
Problematic cannabis use | Administered at Week 1 and Week 20 of CBT for eating disorders.
  Measured using Cannabis Use Disorder Identification Test-Revised. Assesses for indicators of problematic cannabis use, such as inability to reduce use, using in risky circumstances, increased impairment, and frequency of use. Items are answered on a scale of 0 to 4, with higher scores indicating more problematic use. A total score is calculated by summing item scores.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah McComb, Ph.D., C. Psych, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, West 5th Campus, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided